CLINICAL TRIAL: NCT06145321
Title: Continuous Infusion of Granulocyte Colony-stimulating Factor is Associated With an Advantage in Neutrophil Recovery in Hematologic and Oncologic Disorders
Brief Title: Continuous Versus Bolus Administration of G-CSF in Children With Cancer
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Lun Wang, MD, Medical doctor/Clinical physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CVB-1115
Record Dates: First submitted 2023-11-15; First posted 2023-11-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Cancer; Neutropenia; Lenograstim; Filgrastim; G-CSF
Keywords: Pediatric cancer; Neutropenia; G-CSF
MeSH Terms: conditions — Neoplasms; Neutropenia | interventions — Filgrastim; Lenograstim

STUDY DESIGN:
Intervention Model Description: Investigational product(s)：G-CSF (filgrastim) Route of administration: intravenous infusion (with a 5 hours infusion period) or intravenous bolus (with an infusion period of less than one minute)
Who Masked: Participant
Masking Description: We aimed to enroll 40 hospitalized patients in this phase 4 clinical trial. Patients with an ANC lower than 500 cells/mm3 will be randomly categorized into experimental and controlled arms. The experimental arm was designed to receive G-CSF intravenous infusion for 5 hours at a dose of 5 mcg/kg. The controlled arm was designed to receive a G-CSF bolus injection within one minute at a dose of 5 mcg/kg. Three days after treatment initiation, serum white blood cell and differential counts will be followed daily to determine the timing of steady neutrophil recovery. In the following time of another neutropenia event, the experimental arm would cross-switch to the controlled arm and receive corresponding G-CSF according to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental Group (Experimental): G-CSF at a dose of 5 mcg/kg/day intravenously infused for 4 hours
  Interventions: Device: G-CSF administration (bolus injection versus intravenous infusion); Drug: G-CSF administration (bolus injection versus intravenous infusion)
- Control Group (Other): G-CSF at a dose of 5 mcg/kg/day intravenously bolus
  Interventions: Device: G-CSF administration (bolus injection versus intravenous infusion); Drug: G-CSF administration (bolus injection versus intravenous infusion)

INTERVENTIONS:
Device: G-CSF administration (bolus injection versus intravenous infusion) — Route of administration: intravenous infusion (with a 5 hours infusion period) or intravenous bolus (with an infusion period of less than one minute)
  Other Names: Filgrastim, Lenograstim
Drug: G-CSF administration (bolus injection versus intravenous infusion) — Route of administration: intravenous infusion (with a 5 hours infusion period) or intravenous bolus (with an infusion period of less than one minute)
  Other Names: Filgrastim, Lenograstim

SUMMARY:
The investigators hypothesized that in terms of granulocyte colony-stimulating factor (G-CSF) administration, the route of continuous infusion would lead to a faster neutrophil recovery compared to that of bolus administration

DETAILED DESCRIPTION:
The investigators aimed to enroll 40 hospitalized patients in this phase 4 clinical trial. Patients with an ANC lower than 500 cells/mm3 will be randomly categorized into experimental and controlled arms. The experimental arm was designed to receive G-CSF intravenous infusion for 5 hours at a dose of 5 mcg/kg. The controlled arm was designed to receive a G-CSF bolus injection within one minute at a dose of 5 mcg/kg. Three days after treatment initiation, serum white blood cell and differential counts will be followed daily to determine the timing of steady neutrophil recovery. In the following time of another neutropenia event, the experimental arm would cross-switch to the controlled arm and receive corresponding G-CSF according to the study design

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with an age between 0 to 18 years old will be included
* Hematologic and oncologic malignancies

Exclusion Criteria:

* Patients with a diagnosis of myelodysplastic syndrome or severe aplastic anemia will be excluded
* Patients receiving G-CSF treatment 7 days before enrollment will be excluded
* Patients concurrently receiving cytokine therapy or thrombopoietin receptor agonist therapy will be excluded

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Absolute neutrophil counts (ANC) | up to 30 days
  ANC higher than 1500 cells/mm3 for three consecutive days

SECONDARY OUTCOMES:
Hospitalization duration | up to 30 days
  Hospitalization duration from admission to discharge
Re-hospitalization event | up to 5 times
  14 days re-hospitalization event
Clinical sepsis | up to 5 times
  Events of severe bacterial infection during neutropenic period

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Children Hospital, Taoyuan District, ROC, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Detailed informations should be shared if indicated.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: up to one year
Access Criteria: All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB. The formal consent of a subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure. This consent form must be signed by the subject or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.
  Clinical samples will be collected at Chang Gung Medical Foundation. The sequencing data will be stored in the computers of a laboratory with electronic encryption. The clinical and source data can only be assessed by clinical doctors and investigators of the study.

REFERENCES:
- [Result] Theyab A, Algahtani M, Alsharif KF, Hawsawi YM, Alghamdi A, Alghamdi A, Akinwale J. New insight into the mechanism of granulocyte colony-stimulating factor (G-CSF) that induces the mobilization of neutrophils. Hematology. 2021 Dec;26(1):628-636. doi: 10.1080/16078454.2021.1965725. PMID 34494505
- [Result] Dale DC. How I manage children with neutropenia. Br J Haematol. 2017 Aug;178(3):351-363. doi: 10.1111/bjh.14677. Epub 2017 Apr 17. PMID 28419427
- [Result] Blayney DW, Schwartzberg L. Chemotherapy-induced neutropenia and emerging agents for prevention and treatment: A review. Cancer Treat Rev. 2022 Sep;109:102427. doi: 10.1016/j.ctrv.2022.102427. Epub 2022 Jun 21. No abstract available. PMID 35785754
- [Result] Stroncek DF, Matthews CL, Follmann D, Leitman SF. Kinetics of G-CSF-induced granulocyte mobilization in healthy subjects: effects of route of administration and addition of dexamethasone. Transfusion. 2002 May;42(5):597-602. doi: 10.1046/j.1537-2995.2002.00091.x. PMID 12084168
- [Result] Cainap C, Cetean-Gheorghe S, Pop LA, Leucuta DC, Piciu D, Mester A, Vlad C, Ovidiu C, Gherman A, Crisan C, Bereanu A, Balacescu O, Constantin AM, Dicu I, Balacescu L, Stan A, Achimas-Cadariu P, Cainap S. Continuous Intravenous Administration of Granulocyte-Colony-Stimulating Factors-A Breakthrough in the Treatment of Cancer Patients with Febrile Neutropenia. Medicina (Kaunas). 2021 Jun 30;57(7):675. doi: 10.3390/medicina57070675. PMID 34208815
- [Result] de Jong ME, Carbiere T, van den Heuvel-Eibrink MM. The use of an insuflon device for the administration of G-CSF in pediatric cancer patients. Support Care Cancer. 2006 Jan;14(1):98-100. doi: 10.1007/s00520-005-0872-x. Epub 2005 Aug 12. PMID 16096770